CLINICAL TRIAL: NCT05542771
Title: External Validation of the Beta-lactam Target Non-attainment (BATMAN) Risk Score in Adult ICU Patients: a Diagnostic Multivariate Predictive Risk Model
Acronym: BATMAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chantal Kats (Other)
Responsible Party: Sponsor-Investigator, Chantal Kats, MSc Chantal Kats, coordinating researcher (Sponsor is Erasmus Medical Center), Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: NL181245.078.22
Record Dates: First submitted 2022-08-30; First posted 2022-09-15 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Infection, Bacterial; Beta-lactam Antibiotics; Critical Care; Risk Model; Therapeutic Drug Monitoring
Keywords: External validation; Critical care; Risk model; Beta-lactam antibiotics; Therapeutic drug monitoring; infections, bacterial
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4 ml blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intensive care (IC) patients regularly get infections. Sometimes it is even the reason of admission to the intensive care unit. To treat these infections, we give medicines called antibiotics, such as β-lactams antibiotics. Every IC patient receives the same dose of β-lactams antibiotics, while we know this can lead to undertreatment in some IC patients. The BATMAN risk score was created to predict which IC patient is undertreated. This study aims to validate the BATMAN risk score so it can be used in clinical practice.

DETAILED DESCRIPTION:
In order to predict which intensive care unit (ICU) patients are not likely to achieve target attainment of beta-lactam antibiotics, a diagnostic multivariable prediction model was developed using random forest analysis. Gender, age, creatinine, and type of beta-lactam antibiotic were included in the final model and translated into a user-friendly and easy-to-implement risk score. As the name suggests, the beta-lactam target non-attainment (BATMAN) risk score predicts which adult ICU patients fail to achieve target attainment and intents efficient use of TDM of beta-lactam antibiotics. In order to use the BATMAN risk score in as many hospitals as possible in clinical practice, an external validation will be performed by a multicenter prospective observational study. All adult ICU patients admitted to the participating hospitals that are treated with beta-lactam antibiotics will be screened for eligibility. One beta-lactam trough plasma concentration, clinical and non-clinical data will be collected prospectively. To our knowledge, no other beta-lactam target non-attainment risk score for adult ICU patients has yet been developed let alone externally validated. This research is essential because ICU patients are a highly heterogenic group of patients that undergo extensive physiological alterations that will have impact on antibiotic pharmacokinetics, such as beta-lactam antibiotics. For the beta-lactams, achievement of an adequate drug level is associated with a higher likelihood of clinical success and a decrease in the potential for antimicrobial resistance. Yet, target attainment remains a challenge with the traditional 'one-dose-fits-all' strategy.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent has been obtained from the patient or their legally authorised representative
* Age ≥18 years
* Treated with one of the following beta-lactam antibiotics at the ICU with intermitted dosage

  * Amoxicillin (with or without clavulanic acid)
  * Cefotaxime
  * Ceftazidime
  * Cefuroxime
  * Flucloxacillin
  * Meropenem
  * Piperacillin with tazobactam
* Eligible blood material within 36 hours after start of beta-lactam antibiotic to determine target attainment (100%ƒT > MICECOFF).
* Suitable intravenous/intra-arterial access to facilitate sample collection

Exclusion Criteria:

* Pregnancy
* Beta-lactam antibiotic cessation before blood sample collection
* Receiving beta-lactam antibiotic only as prophylaxis within the context of Selective Digestive tract Decontamination (SDD)
* Patients with renal replacement therapy
* Patients with burn injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to the adult general ICU wards and treated with the target antibiotics who meet the inclusion criteria will be included.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Discrimination | Target attainment prediction based on the BATMAN risk score is calculated with patient data within 36 hours after of start therapy. Target attainment based on serum levels are based are measured within 36 hours after start of therapy.
  The discrimination of the diagnostic risk score will be displayed in the concordance index (c-index), which is identical to the area under the receiver operating curve (AUROC), where the true positive rate (y-axis) will be plotted against the false positive rate (x-axis).
Calibration | Target attainment prediction based on the BATMAN risk score is calculated with patient data within 36 hours after of start therapy. Target attainment based on serum levels are based are measured within 36 hours after start of therapy.
  The calibration of the risk score will be assessed with a calibration plot, where the average predicted risk of target non-attainment is compared with the overall event rate of target non-attainment.

OTHER OUTCOMES:
Negative predictive value | Target attainment prediction based on the BATMAN risk score is calculated with patient data within 36 hours after of start therapy. Target attainment based on serum levels are based are measured within 36 hours after start of therapy.
  The ratio of subjects truly diagnosed as negative (target attainment) to all those who had negative test results
Positive predictive value | Target attainment prediction based on the BATMAN risk score is calculated with patient data within 36 hours after of start therapy. Target attainment based on serum levels are based are measured within 36 hours after start of therapy.
  The ratio of subjects truly diagnosed as positive (target non-attainment) to all those who had positive test results.
Sensitivity | Target attainment prediction based on the BATMAN risk score is calculated with patient data within 36 hours after of start therapy. Target attainment based on serum levels are based are measured within 36 hours after start of therapy.
  Sensitivity is the percentage of true positives.
Specificity | Target attainment prediction based on the BATMAN risk score is calculated with patient data within 36 hours after of start therapy. Target attainment based on serum levels are based are measured within 36 hours after start of therapy.
  Specificity is the percentage of true negatives.
Misclassification | Target attainment prediction based on the BATMAN risk score is calculated with patient data within 36 hours after of start therapy. Target attainment based on serum levels are based are measured within 36 hours after start of therapy.
  Percentage of observations that were incorrectly predicted (false negatives and false positives)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Adulla, PhD, Principal Investigator — Erasmus Medical Center
Locations (6):
- Netherlands (6):
  - Isala Hospital, Zwolle, Gelderland
  - VieCuri Medical Center, Venlo, Limburg
  - Erasmus Medical Center, Rotterdam, South Holland
  - Franciscus Gasthuis & Vlietland, Rotterdam, South Holland
  - Haaglanden Medisch Centrum, The Hague, South Holland
  - Diakonessenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to other researchers